CLINICAL TRIAL: NCT03239106
Title: An Open Label Study of Apremilast in Chronic Idiopathic Pruritus
Brief Title: A Study Examining the Medication Apremilast as Treatment for Chronic Itch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-ApremilastCC-10004
Record Dates: First submitted 2017-07-28; First posted 2017-08-03 (Actual); Results first posted 2020-04-20 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Itch
Keywords: itch; pruritus; CIP
MeSH Terms: conditions — Pruritus | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- open label (Experimental): All participants will receive Apremilast 30 mg BID.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg BID daily
  Other Names: Otezla

SUMMARY:
Chronic Itch is a debilitating condition affecting many people. Currently, there are no FDA-approved treatments. Apremilast is an FDA-approved oral medication used to successfully treat the inflammatory skin disorder psoriasis and the inflammatory disorder psoriatic arthritis. This study examines if apremiliast taken twice daily relieves chronic itch.

DETAILED DESCRIPTION:
There is no FDA-approved medication for chronic idiopathic pruritus (CIP). Apremilast has demonstrated notable activity and is approved for treatment in other pruritic inflammatory skin conditions such as psoriasis. The drug is currently being investigated as therapy for atopic dermatitis. Additionally, the investigators have preliminary data to suggest that apremilast's anti-inflammatory properties may work via neuromodulation targeting neuronal cytokine pathways. The proposed study plans to assess the efficacy of apremilast 30 mg BID in the setting of CIP. Durable response to a medication is typically seen within one to two months of starting an efficacious medication in subjects who respond. Therefore, the investigators have designed this study to end at Week 16 to definitively determine efficacy and conclude the study with confidence with regard to both efficacy and failure.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria: A subject who meets all of the following criteria may be included in the study:

* Male and non-pregnant, non-lactating female subjects aged 18 years or older
* Diagnosed with chronic idiopathic pruritus (CIP) with an NRS Itch Score of ≥ 7 at both Screening and Baseline
* Diagnosis of CIP for at least 6 weeks prior to screening
* Willingness to avoid pregnancy or fathering of children
* Ability and willingness to provide written informed consent
* Willing and able to comply with all study requirements and restrictions
* Willing to not participate in any other interventional trial for the duration of their participation
* Subjects must be in good health as determined by medical history, physical examination, electrocardiogram, clinical laboratory tests and vital signs
* Failure of a course 2-week course of treatment with topical triamcinolone 0.1% ointment BID
* Histopathological demonstration of skin eosinophils, mast cell activation, lymphocytic infiltration, and/or dermal edema

Exclusion Criteria:

Key Exclusion Criteria: A subject who meets any of the following criteria will be excluded from the study:

* Chronic pruritus due to a defined primary dermatologic disorder (e.g., atopic dermatitis, psoriasis, etc.)
* Patients with a prior diagnosis of excoriation disorder
* Use of topical treatments for CIP (other than bland emollients) within 1 week of Baseline
* Systemic immunosuppressive or immunomodulating drugs within 4 weeks of Baseline
* Subjects with cytopenias at screening, defined as:

  * Leukocytes < 3 × 109/L.
  * Neutrophils < lower limit of normal.
  * Lymphocytes < 0.5 × 109/L
  * Hemoglobin < 10 g/dL.
  * Platelets < 100 × 109/L.
* Unwilling or unable to follow medication restrictions described in Section 5.6.3, or unwilling or unable to sufficiently washout from use of restricted medication
* Under medical treatment for a skin disease with a therapy listed in the prohibited medications section that may influence the results of the study
* Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal gastrointestinal, endocrine or metabolic dysfunction unless currently controlled and stable, including (but not limited to) the following: Positive for Hepatitis C antibody test (anti-HCF) Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) Positive for HIV (DUO test, p24 antigen)
* Active malignancy
* Active substance abuse or history of substance abuse within 6 months of screening
* History (including family history) or current evidence of congenital long QT syndrome or known acquired QT prolongation
* Exposure to any investigational medication, including placebo, within 60 days of the Baseline Visit
* Subjects who had previously received apremilast
* Subjects with severely impaired liver function (Child-Pugh Class C) or end-stage renal disease on dialysis or at least 1 of the following:

  * Serum creatinine > 1.5 mg/dL
  * Alanine aminotransferase or aspartate aminotransferase ≥ 1.5 × upper limit of normal
* Anyone affiliated with the site or sponsor and/or anyone who may consent under duress
* Any other sound medical reason as determined by the Investigator including any condition which may lead to an unfavorable risk-benefit of study participation, may interfere with study compliance or may confound results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian S. Kim, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Division of Dermatology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: All participants will received apremilast 30 mg PO BID.
Period: Overall Study
Arm/Group | Open Label
Started | 10
Completed | 3
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Key inclusion criteria included age >18 years, diagnosis of chronic pruritus of unknown origin (CPUO) for >6 weeks, Numerical Rating Scale (NRS) itch score of >7, failure of topical triamcinolone 0.1% ointment twice daily (BID) for at least 2 weeks.
Groups:
- Open Label: All participants will receive apremilast 30 mg PO BID.
Arm/Group | Open Label
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
24 hour numerical rating scale (NRS) itch score [Median (Inter-Quartile Range); unit: units on a scale] | 9.25 [7.75 to 10]
1 week NRS itch score [Mean (Standard Deviation); unit: units on a scale] | 8 (0.91)
Dermatology Life Quality Index [Median (Inter-Quartile Range); unit: units on a scale] | 11.5 [8 to 20.5]

OUTCOME MEASURES:

1. Primary Outcome: Absolute NRS Itch Score at Week 16 (End of Treatment)
Description: Participants will complete a Numeric Rating Scale for itch (0 representing "no itching" through 10 representing "worst itch imaginable") will be recalled from prior 24 hours and the prior week.
  0 is the best score (minimum) and 10 is the worst score (maximum) in terms of clinical outcome. This is an ordinal scale that runs from 0 to 10.
Time Frame: Week 16
Population: All patients met criteria for chronic pruritus of unknown origin.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Groups:
- Open Label: All participants will receive apremilast 30 mg PO BID.
  The data were analyzed in an intent-to-treat manner with key primary and secondary endpoints measured as an absolute reduction in NRS itch and DLQI scores, respectively at week 16 from baseline. Thirty percent of the patients completed the study, which did not allow for meaningful intent-to-treat statistical analysis. As an alternative approach, we undertook a LOCF analysis by carrying forward to week 16.
Arm/Group | Open Label
Number analyzed (Participants) | 10
Units on a scale
  24 Hour NRS Itch Score | 7 [1.5 to 10]
  1 Week NRS Itch Score | 7.5 [2 to 9.25]

2. Secondary Outcome: Absolute DLQI at Week 16
Description: Participants will complete a 10 question Dermatology Quality of Life survey at baseline through Week 16
  The DLQI is a numerical scale that scores multiple parameters of skin symptoms on a scale from 0 to 30. 0-1 = no effect at all on a patient's life (most favorable clinical outcome and minimum score), 1-5 = small effect on patient's life, 6-10 = moderate effect on patient's life, 11-20 = very large effect on patient's life, 21-30 = extremely large effect on patient's life (worse clinical outcome and maximum score).
Time Frame: Week 16
Population: Patients who met inclusion criteria with a diagnosis of chronic pruritus of unknown origin
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 10
Score on a scale | 13 [2.5 to 18.75]

3. Secondary Outcome: NRS at Screening, Baseline and Weeks 2,4,8,12,16,and 18
Description: Participants' itch will be measured utilizing the Numeric Rating Scale for itch (0 representing "no itching" through 10 representing "worst itch imaginable") will be recalled from prior 24 hours and the prior week.
  0 is the best score (minimum) and 10 is the worst score (maximum) in terms of clinical outcome. This is an ordinal scale that runs from 0 to 10.
Time Frame: Screening through Week 18 (follow up visit)
Population: Although we started with 10 patients, patients dropped out of the study as it progressed.
Measure: Mean (Standard Deviation); unit: Numerical Rating Scale Itch Score
Arm/Group | Open Label
Number analyzed (Participants) | 10
Numerical Rating Scale Itch Score
  Screening | 8.9 (1.1)
  Baseline (Week 0) | 7.9 (1.6)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 5.7 (3.7)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 6.5 (4.1)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 7.0 (4.2)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 5.7 (5.1)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 3.0 (5.2)
  Week 18: number analyzed (Participants) | 2
  Week 18 | 1.0 (0.0)

4. Secondary Outcome: DLQI at Screening, Baseline, and Weeks 2,4,8,12,16 and 18
Description: Participants will complete a 10 question Dermatology Life Quality Index questionnaire at Screening, Baseline, and Weeks 2,4,8,12,16,18.
Time Frame: Screening through Week 18 (follow up visit)
Population: Although we started with 10 patients, patients dropped out of the study as it progressed.
Measure: Mean (Standard Deviation); unit: Dermatology Life Quality Index Score
Arm/Group | Open Label
Number analyzed (Participants) | 10
Dermatology Life Quality Index Score
  Screening | 15.3 (7.3)
  Baseline (Week 0) | 13.7 (7.6)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 13.3 (9.9)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 10.8 (9.9)
  Week 8: number analyzed (Participants) | 4
  Week 8 | 7.5 (6.5)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 4.7 (6.4)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 2.3 (2.1)
  Week 18: number analyzed (Participants) | 2
  Week 18 | 5.0 (5.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected until the end of the study visit at Week 18 or earlier if the subject dropped out of the study.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=10)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Decreased appetite (General disorders) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the high dropout rate in this study a meaningful intent-to-treat analysis was not possible. Therefore, in addition, we attempted a last observation carried forward (LOCF) analysis as well.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03239106/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03239106/ICF_002.pdf